CLINICAL TRIAL: NCT06251505
Title: Cervical Sagittal Alignment Changes After Correction of Thoracic Adolescent Idiopathic Scoliosis With Severe Thoracic Hypokyphosis: Which Factors Are Predictive? A Multicenter Retrospective Study
Brief Title: Cervical Alignment Changes After Correction of Thoracic Adolescent Idiopathic Scoliosis With Thoracic Hypokyphosis
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Bol-Ter AIS
Record Dates: First submitted 2024-01-15; First posted 2024-02-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: AIS; Cervical Alignment; Thoracic Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The sagittal alignment of Adolescent Idiopathic Scoliosis (AIS) curves has attracted growing interest in recent years, to the extent that it has become a pivotal point in the Lenke classification, with the introduction of a sagittal modifier. In particular, thoracic curves, partly due to the theory of anterior overgrowth, are almost invariably characterized by thoracic hypokyphosis, which can be severe (T5-T12 thoracic kyphosis < 10°, that corresponds to a Lenke - sagittal modifier). However, the development of such a severely abnormal sagittal alignment has consequences that are not limited only to the thoracic region, but it rather results in a disruption of the entire sagittal spinal alignment. In fact, thoracic hypokyphosis tends to shift the C7SVA backward and to decrease the T1 slope. As a compensation, this ultimately leads to the development of a cervical kyphosis in order to translate the head forward and maintain global sagittal balance. While the interplay relationship between thoracic hypokyphosis and the development of cervical kyphosis has been well established in modern literature, the results regarding the amount of spontaneous correction of cervical kyphosis achieved after hypokyphotic AIS correction are conflicting. There are several papers in literature that study the complex relationship between AIS and cervical kyphosis, and they did not report any improvement in cervical lordosis after AIS correction, even when successful restoration of thoracic kyphosis (TK) was achieved. Conversely, other authors did report an improvement in cervical sagittal alignment after AIS correction. The aim of the present paper is firstly to assess the amount of spontaneous change in cervical sagittal alignment after correction of AIS with associated severe thoracic hypokyphosis (<10°). Secondly, the aim of the study is to seek for any radiographical parameter able to predict the postoperative cervical sagittal alignment in these patients, via a multivariate regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* AIS patients with a major thoracic curve (Lenke 1, 2 , 3 patterns), with associated severe thoracic hypokyphosis (TK < 10°; Lenke - modifier) who underwent surgical correction at the participating centers was performed.

Exclusion Criteria:

* Non-idiopathic scoliosis, infantile, juvenile, or adult idiopathic scoliosis diagnosis were considered exclusion criteria

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: AIS patients with a major thoracic curve (Lenke 1, 2 , 3 patterns), with associated severe thoracic hypokyphosis (TK < 10°; Lenke - modifier) who underwent surgical correction at the participating centers was performed.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cervical alignment | 4 years
  to assess the amount of spontaneous change in cervical sagittal alignment after correction of AIS with associated severe thoracic hypokyphosis (<10°)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No